CLINICAL TRIAL: NCT03623087
Title: Combination Chemotherapy Using Cisplatin, Gemcitabine, Ifosfamide, Etoposide, L-asparaginase and Dexamethasone (SIMPLE) for Newly Diagnosed and Relapsed/Refractory NK/T Cell Malignancies
Brief Title: SIMPLE Chemotherapy for NK Lymphoma/Leukaemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yok-lam Kwong, Chair Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-002
Record Dates: First submitted 2018-07-25; First posted 2018-08-09 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Non-Hodgkin's Lymphoma, Relapsed; Non-Hodgkin T-cell Lymphoma; Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Cisplatin; Gemcitabine; Etoposide; Dexamethasone; Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIMPLE (Experimental): cisplatin, gemcitabine, ifosfamide, etoposide (VP-16), L-asparaginase, dexamethasone
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Etoposide (VP-16); Device: Ifosfamide; Drug: Dexamethasone; Drug: L-asparaginase

INTERVENTIONS:
Drug: Cisplatin — SIMPLE
Drug: Gemcitabine — SIMPLE
Drug: Etoposide (VP-16) — SIMPLE
Device: Ifosfamide — SIMPLE
Drug: Dexamethasone — SIMPLE
Drug: L-asparaginase — SIMPLE

SUMMARY:
NK malignancies consist of two different clinical entities, extranodal NK/T cell lymphoma and aggressive NK leukaemia. Queen Mary Hospital (QMH) had started to use PIGLETS chemotherapy for treatment of NK malignancies since 2013, with promising results. The study in QMH had ended because of successful recruitment in the planned number of subjects.

When PIGLETS was used in extranodal NK/T cell lymphoma, patients with stage I/II lymphoma have an overall response rate of nearly 90%, while patients with stage III/IV disease have an overall response rate of around 60%. The figures are comparable to the SMILE chemotherapy previously used. However, PIGLETS regimen carries much lower risk of nephrotoxicity when compared with SMILE. It has since become a standard protocol in management of NK malignancies in our institution.

PIGLETS chemotherapy carries two major problems:

1. the name PIGLETS may appear offensive to some religious populations. (e.g. Muslim)
2. significant nausea/vomiting was seen in previous studies, and these could at least be partially alleviated with substance P antagonist aprepitant

Thus the investigators decided to start a study, renaming the original PIGLETS regimen into SIMPLE chemotherapy, adding aprepitant as antiemetics and to recruit more patients for evaluation of clinical efficacy. The results of SIMPLE chemotherapy will be compared to SMILE in a non-inferiority trial setting.

DETAILED DESCRIPTION:
Natural killer (NK)/T-cell malignancies comprise two related entities, extranodal NK/T cell lymphoma and aggressive NK leukaemia. The disease occurs world-wide but Asian and South American populations are particularly affected, NK/T cell malignancies carry poor prognosis, the response rate is low with conventional CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) or CHOP-like regimen even for newly diagnosed disease. These regimens are typically ineffective for relapsed disease.

In the last 10 years the investigators have employed two different regimen sequentially. The former SMILE regimen (Dexamethasone, methotrexate, ifosfamide, L-asparaginase and etoposide) harness the combination of P-gp independent chemotherapy in management of NK/T cell malignancies with great success. However, nephrotoxicity remained a major concern with the use of this regimen. The SMILE regimen was later modified as PIGLETS regimen (cisplatin, ifosfamide, gemcitabine, L-asparaginase, etoposide, dexamethasone) to reduce the risk of nephrotoxicity while preserving the treatment efficacy. The study with the use of PIGLETS was approved by IRB. The preliminary results of phase II clinical trial with PIGLETS at Queen Mary Hospital resulted in an overall response rate (ORR) of 80% in newly diagnosed disease.

The recruitment was completed with previous PIGLETS phase II trial. The problems with the PIGLETS regimen are:

1. The term 'PIGLETS' may appear to be offensive in some of the ethnicities/religions.
2. Significant nausea and vomiting, which may be delayed after completion of chemotherapy.

In addition, there is a need of further subject recruitment for comparison with SMILE therapy for non-inferiority. In the current study, the regimen was renamed as 'SIMPLE' and aprepitant (a substance P antagonist) was added in the regimen to reduce the incidence of nausea and vomiting. The current study aims to compare SIMPLE to SMILE in a 'non-inferiority' design.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18-80 with biopsy proven extranodal NK/T cell lymphoma, nasal type or aggressive NK leukaemia
2. ECOG performance score <=2

Exclusion Criteria:

1. Poor performance status with ECOG >=3
2. Impairment of renal function (serum creatinine more than or equal to 200umol/L) not otherwise attributed to the tumour involvement.
3. Impairment of liver function with liver parenchymal enzymes 5 times the upper limit of normal range, not otherwise attributed to tumour involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03-14 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by overall response rate measured at the time of best response. | 2 years
  Overall response rate (ORR) is defined as the proportion of patients with reduction in tumor burden of at least 50%.

SECONDARY OUTCOMES:
Adverse events and severe adverse events related to the treatment | 1 year
  Incidence of AE and SAE by severity grading as assessed according to CTCAE v4.03
Progression-free survival (PFS) | 2 years
  PFS is defined as the time from enrolment to progression or death due to any cause. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Overall survival (OS) | 2 years
  OS is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Yok Lam Kwong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided